CLINICAL TRIAL: NCT05976035
Title: Do Taking Supplements Provide Additional Benefits in Rotator Cuff-Related Shoulder Pain?
Brief Title: Exercise vs. Supplements in Rotator Cuff-Related Shoulder Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Aysenur Erekdag, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A-3456789876
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Rotator Cuff Syndrome
Keywords: Exercise; Physical Therapy; Anti-oxidant; Anti-Inflammatory
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Participants will be divided into two groups with equal numbers by computer randomization method.
Who Masked: Outcomes Assessor
Masking Description: The investigator administering the treatment and the investigator performing the assessment will be different. The assessor will not know about the interventions that the participants received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise & Supplement Group (Active Comparator): Exercise & Supplement group will take supplements that are prescribed by the orthopedist every day for 8 weeks in addition to a structured exercise program under the supervision of a physiotherapist 3 days per week for 8 weeks.
  Interventions: Other: Exercise; Other: Supplement
- Exercise Group (Active Comparator): Exercise group will follow a structured exercise program under the supervision of a physiotherapist 3 days per week for 8 weeks.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Structured exercise program under the supervision of a physiotherapist 3 days per week for 8 weeks
Other: Supplement — Receiving supplement that are prescribed by a orthopedist every day for 8 weeks
  Arms: Exercise & Supplement Group

SUMMARY:
Rotator cuff-related shoulder pain is a pathology characterized by pain and functional impairment originating from one or more rotator cuff tendons. The lifetime incidence of rotator cuff-related shoulder pain is around 67%, with an annual incidence exceeding 1%. Many patients continue to experience pain and functional loss for up to one year, and more than half of the patients report shoulder pain persisting for over three years.

The pathophysiology underlying rotator cuff-related shoulder pain continues to be a subject of ongoing research and uncertainty, with many aspects yet to be fully elucidated. The most common belief regarding its pathogenesis involves the role of inflammation. This hypothesis is supported by the accumulation of inflammatory cells in tendons, oxidative stress, and increased levels of pro-inflammatory cytokines. In tendon pathologies with inflammatory cell accumulation and increased cytokine levels, the use of antioxidants and anti-inflammatory agents in addition to conservative treatment contributes to tendon healing. Anti-oxidants and anti-inflammatories are substances capable of preventing or delaying certain cell damage.The use of anti-inflammatory and antioxidant supplements such as Vitamin C (Vit-C), Vitamin D (Vit-D), Omega-3, and Magnesium (Mg) is recommended. Despite indicating exercise as the gold standard for managing rotator cuff-related shoulder pain and the demonstrated anti-inflammatory and anti-oxidant properties of the mentioned supplements, there are still gaps in the understanding of their effectiveness in rotator cuff-related shoulder pain.

Based on these gaps, the goal of this study is to investigate the effects of supplements (Vit-C, Vit-D, Omega-3, and Mg) given in addition to exercise on patients' blood parameters (TNF-a, IL-6, and CRP levels), pain, functional status, quality of life, and patient satisfaction in individuals with rotator cuff-related shoulder pain.

DETAILED DESCRIPTION:
58 participants older than 40 years of age with rotator cuff-related shoulder pain for at least 3 months will be included in the study. Signed voluntary consent will be obtained from the patients. Participants will be divided into two groups. Study groups will be as follows: a) Exercise & Supplement Group and b) Exercise Group.

ELIGIBILITY:
Inclusion Criteria:

* Being over the age of 40
* Diagnosing with rotator cuff-related shoulder pain confirming through clinical examination (Hawkins Kennedy and Empty Can tests) and MRI imaging
* Having shoulder pain for at least three months

Exclusion Criteria:

* Having full-thickness or massive rotator cuff tear,
* Having a history of symptoms onset due to trauma,
* Having a history of surgery on the same shoulder,
* Having shoulder passive external rotation <30° and flexion <120°,
* Having shoulder instability,
* Having an allergy to any supplement,
* Having psychological, emotional, or cognitive problems
* Presence of shoulder problems caused by systemic diseases,
* Presence of diabetes, presence of pregnancy or breastfeeding,
* Malignancy.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | change from baseline pain at 12 weeks
  The scale has range 0 to 10mm. The left side (0mm) shows no pain, and the right side (10mm) shows the most severe pain imaginable. Patients will be asked to mark the severity of their shoulder pain at a point on the scale using this scale. Higher points indicate higher severity and lower points indicate lower severity.
The American Shoulder and Elbow Surgeons Standardized Shoulder Assessment (ASES) | change from baseline pain at 12 weeks
  Among the self-assessment of the patients, there are 11 items including pain level and functionality. For pain in scoring, they describe pain of increasing severity between 0 and 10; In functionality, a 4-point Likert-type scale is used to determine whether they can perform activities of daily living or not. The total score ranges from 0 (absence of function) to 100 (normal function).
Quick Disabilities of The Arm, Shoulder and Hand Questionnaire (Quick DASH) | change from baseline pain at 12 weeks
  Quick DASH is an 11-item questionnaire used to assess upper extremity functionality. The score ranges from 0 (no injury) to 100 (most severe injury).

SECONDARY OUTCOMES:
Rotator Cuff Quality of Life (RC-QoL) | 3 times for 12 weeks
  It is a self-assessment questionnaire consisting of a total of 34 questions and 5 sections assessing the disease-specific quality of life. Each question is assessed on a 100 mm visual analog scale, with 0 representing the lowest score and 100 the best score, and the total score is given as a percentage. Low scores represent low quality of life.
Global Rating of Change Scale (GRC) | 3 times for 12 weeks
  It is a scale to evaluate patient satisfaction. It is designed to determine the extent to which the patient improves or worsens over time. In our study, the change between the pre-treatment status of the participants and their current status at the 8th and 12th weeks after the treatment will be questioned. In our study, GRC consisting of 5 levels between -2 and +2 value ranges (-2: I am much worse, -1: I am worse, 0: I am the same, 1: I am better, 2: I am much better) will be preferred.

CONTACTS AND LOCATIONS:
Overall Officials: Derya Çelik, Prof., Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Department of Physical Therapy and Rehabilitation, Faculty of Health Sciences, Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Lewis J, McCreesh K, Roy JS, Ginn K. Rotator Cuff Tendinopathy: Navigating the Diagnosis-Management Conundrum. J Orthop Sports Phys Ther. 2015 Nov;45(11):923-37. doi: 10.2519/jospt.2015.5941. Epub 2015 Sep 21. PMID 26390274
- [Background] Luime JJ, Koes BW, Hendriksen IJ, Burdorf A, Verhagen AP, Miedema HS, Verhaar JA. Prevalence and incidence of shoulder pain in the general population; a systematic review. Scand J Rheumatol. 2004;33(2):73-81. doi: 10.1080/03009740310004667. PMID 15163107
- [Background] Tashjian RZ. Epidemiology, natural history, and indications for treatment of rotator cuff tears. Clin Sports Med. 2012 Oct;31(4):589-604. doi: 10.1016/j.csm.2012.07.001. Epub 2012 Aug 30. PMID 23040548
- [Background] Macfarlane GJ, Hunt IM, Silman AJ. Predictors of chronic shoulder pain: a population based prospective study. J Rheumatol. 1998 Aug;25(8):1612-5. PMID 9712108
- [Background] Litchfield R. Progressive strengthening exercises for subacromial impingement syndrome. Clin J Sport Med. 2013 Jan;23(1):86-7. doi: 10.1097/JSM.0b013e31827e9fb5. PMID 23269329
- [Background] Vaysman M, Alben M, Todd M, Ruotolo C. Pharmacologic Enhancement of Rotator Cuff Repair: A Narrative Review. Orthop Rev (Pavia). 2022 Sep 4;14(3):37782. doi: 10.52965/001c.37782. eCollection 2022. PMID 36072503
- [Background] Yuan T, Qian H, Yu X, Meng J, Lai CT, Jiang H, Zhao JN, Bao NR. Proteomic analysis reveals rotator cuff injury caused by oxidative stress. Ther Adv Chronic Dis. 2021 Mar 17;12:2040622320987057. doi: 10.1177/2040622320987057. eCollection 2021. PMID 33796243
- [Background] Metsios GS, Moe RH, Kitas GD. Exercise and inflammation. Best Pract Res Clin Rheumatol. 2020 Apr;34(2):101504. doi: 10.1016/j.berh.2020.101504. Epub 2020 Apr 2. PMID 32249021
- [Background] Delgado DA, Lambert BS, Boutris N, McCulloch PC, Robbins AB, Moreno MR, Harris JD. Validation of Digital Visual Analog Scale Pain Scoring With a Traditional Paper-based Visual Analog Scale in Adults. J Am Acad Orthop Surg Glob Res Rev. 2018 Mar 23;2(3):e088. doi: 10.5435/JAAOSGlobal-D-17-00088. eCollection 2018 Mar. PMID 30211382
- [Background] Celik D, Atalar AC, Demirhan M, Dirican A. Translation, cultural adaptation, validity and reliability of the Turkish ASES questionnaire. Knee Surg Sports Traumatol Arthrosc. 2013 Sep;21(9):2184-9. doi: 10.1007/s00167-012-2183-3. Epub 2012 Aug 30. PMID 22932692
- [Background] Beaton DE, Wright JG, Katz JN; Upper Extremity Collaborative Group. Development of the QuickDASH: comparison of three item-reduction approaches. J Bone Joint Surg Am. 2005 May;87(5):1038-46. doi: 10.2106/JBJS.D.02060. PMID 15866967
- [Background] Cinar-Medeni O, Ozengin N, Baltaci G, Duzgun I. Turkish version of the Rotator Cuff Quality of Life questionnaire in rotator cuff-impaired patients. Knee Surg Sports Traumatol Arthrosc. 2015 Feb;23(2):591-5. doi: 10.1007/s00167-014-3290-0. Epub 2014 Sep 11. PMID 25209207
- [Background] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623
- [Background] Matthews TJ, Hand GC, Rees JL, Athanasou NA, Carr AJ. Pathology of the torn rotator cuff tendon. Reduction in potential for repair as tear size increases. J Bone Joint Surg Br. 2006 Apr;88(4):489-95. doi: 10.1302/0301-620X.88B4.16845. PMID 16567784
- [Background] Millar NL, Hueber AJ, Reilly JH, Xu Y, Fazzi UG, Murrell GA, McInnes IB. Inflammation is present in early human tendinopathy. Am J Sports Med. 2010 Oct;38(10):2085-91. doi: 10.1177/0363546510372613. Epub 2010 Jul 1. PMID 20595553
- [Background] Andersson G, Backman LJ, Scott A, Lorentzon R, Forsgren S, Danielson P. Substance P accelerates hypercellularity and angiogenesis in tendon tissue and enhances paratendinitis in response to Achilles tendon overuse in a tendinopathy model. Br J Sports Med. 2011 Oct;45(13):1017-22. doi: 10.1136/bjsm.2010.082750. Epub 2011 May 2. PMID 21540192